CLINICAL TRIAL: NCT06369077
Title: Cross-over Comparison of Latanoprost QOD With Dor-tim QAM to Tim-brim-dor-bim(Atoprost) qd or Lat QD With Dor-tim BID
Brief Title: How Much Does Reduced Dosing of Latanoprost and Dorzolamide-timolol Affect Pressure?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The 95% confidence interval for non-inferiority was met before planned enrollment was reached.
Sponsor: CT Glaucoma Associates (Other)
Responsible Party: Principal Investigator, Peter E. Libre, Medical Director, CT Glaucoma Associates
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTGlaucoma1
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma, Open-Angle; Glaucoma; Drugs
Keywords: dosing
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — dorzolamide-timolol combination; Latanoprost; Timolol

STUDY DESIGN:
Intervention Model Description: Subjects will have baseline IOP measurements (7-9 am and 3-5 pm) after using using latanoprost every other day and dorzolamide-timolol every morning. They will then randomly be assigned in phase 2 to either: double the frequency to latanoprost daily and dorzolamide-timolol twice daily; or use every morning compounded timolol-brimonidine-dorzolamide-bimatoprost. IOP measurements will be repeated 3 weeks after using the phase 2 medications. For phase 3, subjects will use the treatment to which they were not assigned in phase 2, and IOP measurements will again be repeated 3 weeks later.
  At each study visit, dry eye signs will be assessed and brief dry eye survey will be administered.
Who Masked: Outcomes Assessor
Masking Description: Technician measuring IOP and assessing dry eye is masked regarding phase 2 and phase 3 crossover assignment order.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- full dose lat dor-tim; tim-brim-dor-bim (Active Comparator): After baseline IOP measurements, subjects in this arm will use the full dose full dose latanoprost and dorzolamide-timolol in phase 2, and then timolol-brimonidine-dorzolamide-bimatoprost in phase 3.
  Interventions: Drug: dorzolamide/timolol
- tim-brim-dor-bim; full dose lat dor-tim (Active Comparator): After baseline IOP measurements, subjects in this arm will use timolol-brimonidine-dorzolamide-bimatoprost in phase 2, and then full dose latanoprost and dorzolamide-timolol in phase 3.
  Interventions: Drug: dorzolamide/timolol

INTERVENTIONS:
Drug: dorzolamide/timolol — Compare half-frequency dosing of latanoprost and dorzolamide/timolol to full dosing. Compare also to timolol/brimonidine/dorzolamide/bimatoprost
  Other Names: latanoprost; timolol/brimonidine/dorzolamide/bimatoprost

SUMMARY:
IOP effect of half-dose latanoprost dorzolamide-timolol will be compared to full dose. Further comparison will be made timolol-brimonidine-dorzolamide-bimatoprost. Dry eye effects of the different treatments will be assessed.

DETAILED DESCRIPTION:
Subjects will have baseline IOP measurements (7-9 am and 3-5 pm) after using using latanoprost every other day and dorzolamide-timolol every morning. They will then randomly be assigned in phase 2 to either: double the frequency to latanoprost daily and dorzolamide-timolol twice daily; or use every morning compounded timolol-brimonidine-dorzolamide-bimatoprost. IOP measurements will be repeated 3 weeks after using the phase 2 medications. For phase 3, subjects will use the treatment to which they were not assigned in phase 2, and IOP measurements will again be repeated 3 weeks later.

At each study visit, dry eye signs will be assessed and brief dry eye survey will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult glaucoma patients who are taking drops: dor-tim and Latanoprost Ophthalmic Solution 0.005% (Lat) and come in for an appointment during the trial period

Exclusion Criteria:

* Patients who had an SLT or glaucoma procedure or surgery within 3 months of enrollment will be excluded. Other exclusion criteria include the logistical inability to follow up with the trial, the inability to relax eye muscles for an accurate tonometry measurement, and the inability to instill medications.

The final determination to be included in the study will be made by the Physician on the day of the appointment.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | 3 weeks after each phase
  measured by pneumatonometry and Goldmann tonometry

SECONDARY OUTCOMES:
dry eye | 3 weeks after each phase
  assess punctate staining of cornea and subjective symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Libre, MD, Principal Investigator — CT Glaucoma Associates
Locations (1):
- CT Glaucoma Associates, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No